CLINICAL TRIAL: NCT04278196
Title: Computer Assisted Quality-monitoring for Magnet-controlled Capsule Endoscopy: a Prospective Case-control Study.
Status: Completed | Type: Observational
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Vice President of Qilu Hospital, Shandong University
Other Study IDs: 2020SDU-QILU-24
Record Dates: First submitted 2020-02-19; First posted 2020-02-20 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Magnet Controlled Capsule Endoscopy
Keywords: Artificial intelligence; Magnet controlled capsule endoscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: AI-Box — AI-box is a system fixed adjacent to magnet controlled capsule endoscopy. Patients who accept the check of magnet controlled capsule endoscopywill be enrolled .

SUMMARY:
During the past several years，MCE（magnet controlled endoscopy）has made great process in detecting lesions of gastric as well as screening. Compared with conventional endoscopy, magnetically controlled capsule endoscopy can be further optimized in gastric examination. So we make an AI for operators to help improve the quality of MCE and record the mucosa visibilty of gastirc.

DETAILED DESCRIPTION:
We developed a new artificial intelligence for quality improving during the operation of magnet controlled endoscopy. The AI can help operators screen every part of gastric and then evaluate the visibilty of gastic. Also, It can be record time of the opration. Other than that ,we compared the performancce of AI with experts.

ELIGIBILITY:
Inclusion Criteria:

* patients between 18 and75
* patients who can sign informed consent

Exclusion Criteria:

* patients who are unsuitable to accept the check

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patients who acccept the magnet controlled capsule endoscopy with the help of "AI-box"will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
The integrity of the magnet controlled capsule endoscopy | 2 months
  The performance of the operator developing the MCE in screen the gastric without omissions
The visibilty of the gastric | 2 months
  Evaluating the performance of AI to recognize the visibility of gastric mucosa
The time of operation in gastric | 2 months
  Calculating the time of the magnet controlled capsule endoscapy

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gastroenterology, Qilu Hospital, Shandong University, Jinan, Shandong, China